CLINICAL TRIAL: NCT01238263
Title: Autologous Serum Skin Testing in Patients With Atopic Dermatitis Autologous Serum Skin Testing in Patients With Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Silvan State Hospital, Dermatology department
Other Study IDs: yavuzyesilova
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2009-05

CONDITIONS: Atopic Dermatitis, Serum Skin Test
Keywords: Atopic dermatitis, autologous serum skin testing, IgE autoantibodies
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Recently, IgE-type autoantibodies against self proteins have been detected in the serum of the atopic dermatitis patients. The role of this IgE autoantibodies involved in the pathogenesis of atopic dermatitis is not known, yet. But, there may be a correlation between the severity of the disease and the serum levels of this autoantibodies. The autologous serum skin testing is applied to both atopic dermatitis patients and healthy control and the results are estimated in this study.The investigators detected 70% positive autologous serum skin testing in atopic dermatitis patients and test positivity was higher in patients with atopy history, moderately severe disease calculated by SCORAD index and high serum IgE levels.

ELIGIBILITY:
Inclusion Criteria:

* Sixty AD patients and 30 healthy individuals

Exclusion Criteria:

* . The patients showing evidence of any other disease are not included to our study. No drug was allowed fourteen days prior to the test, including antihistamines and steroids.

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 90
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)